CLINICAL TRIAL: NCT04484649
Title: Development and Pilot Testing of Sleeping Healthy/Living Healthy, a Comprehensive Sleep Intervention for Adolescents in Urban School Based Health Center (SBHCs): Phase II or Randomized Pilot Trial
Brief Title: Sleeping Healthy/Living Healthy Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAS9595
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Sleep; Psychological Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Sleeping Healthy/Living Healthy
  Interventions: Behavioral: Sleeping Healthy/Living Healthy
- Control (Active Comparator): Attention Control
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Sleeping Healthy/Living Healthy — Sleeping Healthy/Living Healthy will be a school based health center (SBHC)-based intervention integrating mind-body integrative health (MBIH) and sleep hygiene strategies to improve sleep quality in urban adolescents. The Sleeping Healthy/Living Healthy intervention content and format will be determined in a Development Phase 1. The investigator anticipates the intervention will consist of two group and two one-on-one sessions. The intervention will be grounded in social-cognitive theory and use motivational interviewing to support MBIH and sleep hygiene strategies. Sessions will be delivered once per week by SBHC providers and health educators.
  Arms: Intervention
Behavioral: Attention Control — The Attention Control Intervention condition will meet the requirements for a comparison treatment for testing behavioral interventions - equivalent in contact time, credible and interesting, and exert limited treatment effects.
  In the same number of sessions and format as the Sleeping Healthy/Living Healthy intervention (anticipated to be two group and two one-on-one sessions delivered once per week by SBHC providers and health educators), the study will teach participants about sleep and other health topics relevant to adolescents (e.g., nutrition, injury prevention) devoid of the MBIH elements in our integrated intervention.
  Arms: Control

SUMMARY:
This pilot study will: (1) develop Sleeping Healthy/Living Healthy, a school-based health center (SBHC) intervention that combines MBIH and sleep hygiene strategies to improve sleep quality in urban adolescents with poor sleep quality; (2) evaluate the feasibility and acceptability of intervention procedures; and (3) assess the preliminary intervention effects on sleep quality in urban adolescents.

This study includes a development phase and a pilot individually-randomized group treatment (IRGT) phase. In Year 1, the investigators will develop the novel integrated intervention using an iterative participatory design process. In Year 2, the investigators will conduct an IRGT trial with 60 adolescents with insufficient sleep recruited from two SBHCs in New York City. Adolescents will be randomized 1:1 to receive the intervention or an attention control of equal intensity and duration. Process evaluation interviews guided by a rigorous fidelity framework with adolescents and with SBHC providers and personnel will be conducted to obtain feedback regarding intervention procedures.

DETAILED DESCRIPTION:
Poor sleep quality, which contributes to impaired functioning, is elevated in urban, ethnic/racial minority adolescents due, in part, to poor sleep hygiene. Despite successful sleep hygiene interventions in younger children, none focus on adolescents, a group with unique developmental needs. Urban adolescents face unique contextual stressors, which may contribute to ineffective use of sleep hygiene behaviors. Mind-body integrative (MBIH) approaches (e.g. yoga, meditation) improve sleep quality in adults, but are rarely applied to adolescents. MBIH has been shown to reduce stress among adolescents. Taken together, this suggests that integrating MBIH with sleep hygiene strategies has the potential for a synergistic effect on improving sleep quality, yet no interventions concurrently use MBIH and sleep hygiene with adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 13.0 -17.9;
* Grade 9 - 11;
* Currently enrolled as a patient in one of the participating SBHCs; and
* Report sleep duration < 8 hours (below the minimally recommended number of hours of sleep for this age group through the following questions: What time do you: a) usually fall asleep on weekdays and b) usually wake up on weekdays?).

Exclusion Criteria:

* Report of prior diagnosis of a sleep disorder, such as sleep disordered breathing, restless leg syndrome, or periodic limb movement;
* Significant developmental delay and/or severe psychiatric or medical conditions that preclude completion of study procedures or confound analyses; or
* Not capable of communicating (reading, speaking, writing) in English.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Garbers-Adams, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Attention Control
  Attention Control: The Attention Control Intervention condition will meet the requirements for a comparison treatment for testing behavioral interventions - equivalent in contact time, credible and interesting, and exert limited treatment effects.
  In the same number of sessions and format as the Sleeping Healthy/Living Healthy intervention (anticipated to be two group and two one-on-one sessions delivered once per week by SBHC providers and health educators), the study will teach participants about sleep and other health topics relevant to adolescents (e.g., nutrition, injury prevention) devoid of the MBIH elements in our integrated intervention.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 30 | 31
Completed (Completed at least 1 day of actigraphy post intervention) | 22 | 26
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Did not submit actigraphy post interc\vention | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Customized [Number; unit: years]
  14 years | 3 | 3 | 6
  15 years | 8 | 11 | 19
  16 years | 10 | 11 | 21
  17 years | 9 | 6 | 15
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 10 | 10 | 20
  Preferred not to answer | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 27 | 51
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Average Sleep Duration (Past 2 Weeks)
Description: Measured using actigraphy. Measured in minutes.
Time Frame: Baseline (Day 0)
Population: Only 27 out of 30 Control and 27 out of 31 Intervention participants completed the actigraphy and were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Intervention
Number analyzed (Participants) | 27 | 27
minutes | 404.2418126 (41.4605752) | 394.9457195 (54.7797086)

2. Primary Outcome: Average Sleep Duration (Past 2 Weeks)
Description: Measured with actigraphy. Measured in minutes.
Time Frame: Immediate Post (up to 7 weeks after baseline)
Population: Only 18 out of 30 Control and 24 out of 31 Intervention participants completed the actigraphy and were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Intervention
Number analyzed (Participants) | 18 | 24
minutes | 419.5089676 (57.9706010) | 399.1041454 (49.9715607)

3. Primary Outcome: Average Sleep Duration (Past 2 Weeks)
Description: Measured in actigraphy. Measured in minutes.
Time Frame: Follow-up (up to 2.5 months)
Population: Only 19 out of 30 Control and 18 out of 31 Intervention participants completed the actigraphy and were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 18
minutes | 408.5679825 (35.9948487) | 395.8340439 (50.3787645)

4. Primary Outcome: Sleep Fragmentation - Sleep Efficiency (%) (Past Month)
Description: Represented as a percentage. Sleep efficiency = (# hours slept/# hours in bed) X 100% Sleep efficiency can range from 0-100%, with higher sleep efficiency representing better sleep.
  The numerator and denominator will be measured through actigraphy.
Time Frame: Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Arm/Group | Control | Intervention
Number analyzed (Participants) | 27 | 27
percentage of sleep efficiency | 88.7501893 (3.2706091) | 87.1876309 (3.9030391)

5. Primary Outcome: Sleep Fragmentation - Sleep Efficiency (%) (Past Month)
Description: as for outcome 4
Time Frame: Immediate Post (up to 7 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Arm/Group | Control | Intervention
Number analyzed (Participants) | 18 | 24
percentage of sleep efficiency | 88.5538488 (6.4652919) | 87.8333318 (4.1461175)

6. Primary Outcome: Sleep Fragmentation - Sleep Efficiency (%) (Past Month)
Description: as for outcome 4
Time Frame: Follow-up (up to 2.5 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 18
percentage of sleep efficiency | 89.2803736 (3.1858765) | 88.4959747 (3.6605489)

7. Primary Outcome: Sleep Fragmentation - Number of Sleep Disruptions (Past Month)
Description: Number of sleep disruptions (number of times awakened) per night (mean, in past month): measured using actigraphy.
Time Frame: Baseline (Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of times awakened
Arm/Group | Control | Intervention
Number analyzed (Participants) | 27 | 27
number of times awakened | 32.3090725 (7.3284517) | 36.1768219 (8.5199704)

8. Primary Outcome: Sleep Fragmentation - Number of Sleep Disruptions (Past Month)
Description: Number of sleep disruptions (number of times awakened) per night (mean, in past month): measured using actigraphy.
Time Frame: Immediate Post (up to 7 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of times awakened
Arm/Group | Control | Intervention
Number analyzed (Participants) | 18 | 24
number of times awakened | 33.6921279 (9.9379062) | 35.9452319 (11.2391805)

9. Primary Outcome: Sleep Fragmentation - Number of Sleep Disruptions (Past Month)
Description: Number of sleep disruptions (number of times awakened) per night (mean, in past month): measured using actigraphy.
Time Frame: Follow-up (up to 2.5 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of times awakened
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 18
number of times awakened | 33.7649958 (10.3250768) | 32.9682422 (10.0477777)

10. Secondary Outcome: Score on Pittsburgh Sleep Quality Index (PSQI Global Score)
Description: Subjective sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), which contains 19 self-rated questions. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Error); unit: global score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
global score on a scale | 7.73 (2.90) | 8.48 (2.98)

11. Secondary Outcome: Score on Pittsburgh Sleep Quality Index (PSQI Global Score)
Description: as for outcome 10
Time Frame: Immediate Post (up to 7 weeks after baseline)
Measure: Mean (Standard Error); unit: global score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
global score on a scale | 6.44 (3.06) | 5.07 (2.24)

12. Secondary Outcome: Score on Pittsburgh Sleep Quality Index (PSQI Global Score)
Description: as for outcome 10
Time Frame: Follow-up (up to 2.5 months)
Measure: Mean (Standard Error); unit: global score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
global score on a scale | 6.07 (2.02) | 4.59 (2.44)

13. Secondary Outcome: Score on the Perceived Stress Scale (PSS)
Description: Stress will be measured using Perceived Stress Scale (past month). The PSS has 10 items, completed using self-report. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress; scores ranging from 14-26 would be considered moderate stress; scores ranging from 27-40 would be considered high perceived stress.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
score on a scale | 28.50 (5.26) | 29.07 (6.11)

14. Secondary Outcome: Score on the Perceived Stress Scale (PSS)
Description: as for outcome 13
Time Frame: Immediate Post (up to 7 weeks after baseline)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
score on a scale | 29.04 (6.23) | 27.11 (5.61)

15. Secondary Outcome: Score on the Perceived Stress Scale (PSS)
Description: as for outcome 13
Time Frame: Follow-up (up to 2.5 months)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
score on a scale | 28.64 (6.71) | 26.07 (6.14)

16. Secondary Outcome: Score on the PROMIS Psychological Stress Experiences Survey - T Score
Description: Stress will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Psychological Stress Experiences Ped Short Form (SF) v1.0 (past 7 days), an 8-item self report. For PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. A higher PROMIS T-score represents more of the concept being measured. For the Psychological Stress Experiences, a T-score of 60 is one standard deviation (SD) worse than average.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 61.74 (8.68) | 62.12 (9.98)

17. Secondary Outcome: Score on the PROMIS Psychological Stress Experiences Survey - T Score
Description: as for outcome 16
Time Frame: Immediate Post (up to 7 weeks after baseline)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 58.70 (9.45) | 57.46 (7.97)

18. Secondary Outcome: Score on the PROMIS Psychological Stress Experiences Survey - T Score
Description: as for outcome 16
Time Frame: Follow-up (up to 2.5 months)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 59.15 (8.36) | 57.83 (11.82)

19. Secondary Outcome: Score on the PROMIS Pediatric Anxiety Short Form 8a v2.0 - T-Score
Description: Anxiety will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Anxiety Short Form 8a v2.0, an 8-item questionnaire assessing self-reported fear, anxious misery, and hyperarousal. Using a five-point frequency scale, ranging from 1 (never) to 5 (almost always), adolescents indicate how frequently or infrequently they felt various dimensions of anxiety (e.g., nervous, scared, worried) in the past 7 days. PROMIS instruments are scored using item-level calibrations.
  For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. A higher PROMIS T-score represents more of the concept being measured. For the Pediatric Anxiety, a T-score of 60 is one standard deviation (SD) worse than average.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 52.82 (7.79) | 53.63 (12.13)

20. Secondary Outcome: Score on the PROMIS Pediatric Anxiety Short Form 8a v2.0 - T Score
Description: as for outcome 19
Time Frame: Immediate Post (up to 7 weeks after baseline)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 50.15 (9.26) | 50.17 (8.88)

21. Secondary Outcome: Score on the PROMIS Pediatric Anxiety Short Form 8a v2.0 - T Score
Description: as for outcome 19
Time Frame: Follow-up (up to 2.5 months)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 51.79 (7.89) | 51.48 (11.02)

22. Secondary Outcome: Score on the PROMIS Pediatric Sleep-Related Impairment Short Form 8a v1.0 - T Score
Description: Subjective sleep-related impairment will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Sleep-Related Impairment Short Form 8a v1.0, an 8-item questionnaire focusing on self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Adolescents rate various aspects of their sleep over the past 7 days on a 5-point frequency scale ranging from 1 (never) to 5 (always). PROMIS instruments are scored using item-level calibrations.
  For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For the Pediatric Sleep-Related Impairment, a T-score of 60 is one standard deviation (SD)
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 61.71 (7.78) | 91.43 (168.67)

23. Secondary Outcome: Score on the PROMIS Pediatric Sleep-Related Impairment Short Form 8a v1.0 - T Score
Description: Subjective sleep-related impairment will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Sleep-Related Impairment Short Form 8a v1.0, an 8-item questionnaire focusing on self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Adolescents rate various aspects of their sleep over the past 7 days on a 5-point frequency scale ranging from 1 (never) to 5 (always). PROMIS instruments are scored using item-level calibrations.
  For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For the Pediatric Sleep-Related Impairment, a T-score of 60 is one standard deviation (SD) worse than average.
Time Frame: Immediate Post (up to 7 weeks after baseline)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 60.08 (8.01) | 55.09 (7.65)

24. Secondary Outcome: Score on the PROMIS Pediatric Sleep-Related Impairment Short Form 8a v1.0 - T Score
Description: as for outcome 23
Time Frame: Follow-up (up to 2.5 months)
Measure: Mean (Standard Error); unit: PROMIS T-score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
PROMIS T-score on a scale | 59.68 (7.90) | 53.22 (10.32)

25. Secondary Outcome: Score on MAAS-A (Mindfulness Attention Awareness Scale - Adolescents)
Description: Mindfulness will be measured using the MAAS-A, a self-reported 14-item questionnaire that measures the level of mindfulness, defined as "a receptive state of attention that, informed by an awareness of present experience, simply observes what is taking place." The MAAS-A is an adapted adolescent version of the validated Mindful Attention Awareness Scale (MAAS), which was developed for use with adult populations and considers mindfulness to be a one-dimensional construct. Using a six-point scale, ranging from 1 (almost always) to 6 (almost never), adolescents indicate how frequently or infrequently they currently have each experience. The score is the mean of the 14 items with higher scores reflecting higher trait mindfulness.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
score on a scale | 3.73 (1.10) | 3.70 (1.12)

26. Secondary Outcome: Score on MAAS-A (Mindfulness Attention Awareness Scale - Adolescents)
Description: as for outcome 25
Time Frame: Immediate Post (up to 7 weeks after baseline)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
score on a scale | 4.04 (1.11) | 4.23 (0.92)

27. Secondary Outcome: Score on MAAS-A (Mindfulness Attention Awareness Scale - Adolescents)
Description: as for outcome 25
Time Frame: Follow-up (up to 2.5 months)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 31
score on a scale | 4.05 (1.11) | 4.45 (1.05)

ADVERSE EVENTS:
Time Frame: Up to 2.5 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04484649/Prot_SAP_000.pdf